CLINICAL TRIAL: NCT06005571
Title: Effect of Silane Coupling Treatment on the Clinical Performance of Direct Repaired Resin-based Composite: A Randomized Controlled Trial.
Brief Title: Effect of Silane Coupling on the Clinical Performance of Repaired Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zakereyya Albashaireh, Professor of restorative dentistry, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220082
Record Dates: First submitted 2023-06-18; First posted 2023-08-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Defective Composite Restorations
Keywords: Silane; Sandblasting of tooth surfaces; Clinical trial; dentine bonding; Composite repair; defective restorations
MeSH Terms: interventions — Adhesives

STUDY DESIGN:
Intervention Model Description: Three groups of patients were randomly assigned to three different treatment protocols of defective composite restoration repair.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients who participated in the study and the assessor of the treatment outcome did not know the type of treatment procedure received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control: traditional acid etch treatment group (Active Comparator): Traditional acid etching to the tooth and old restoration surfaces and then adhesive application.
  Interventions: Procedure: composite restoration repair by traditional acid etch treatment procedure and adhesive.
- Silane-Adhesive treatment group (Experimental): Acid cid etching of prepared tooth tissues and old restoration surfaces, silane solution application, and then adhesive application.
  Interventions: Procedure: Composite restoration repair by acid etching, silane solution application, and then adhesive.
- Sandblast-Silane-Adhesive treatment group (Experimental): First sandblasting the old composite filling surfaces, then acid etching of prepared tooth tissues the restoration, then silane application followed by adhesive application.
  Interventions: Procedure: Composite restoration repair by sandblasting first, then acid etching, silane solution application, and then adhesive.

INTERVENTIONS:
Procedure: composite restoration repair by traditional acid etch treatment procedure and adhesive. — Recurrent caries surrounding the defective restoration was removed and the surfaces were coditoned with acid and adhesive then new repair composite was addded to repair the old restoration and restore the carious cavity.
  Arms: Control: traditional acid etch treatment group
Procedure: Composite restoration repair by acid etching, silane solution application, and then adhesive. — Recurrent caries surrounding the defective restoration was removed and the surfaces were coditoned with acid, then silane applied, next adhesive then new repair composite was addded to repair the old restoration and restore the carious cavity.
  Arms: Silane-Adhesive treatment group
Procedure: Composite restoration repair by sandblasting first, then acid etching, silane solution application, and then adhesive. — Recurrent caries surrounding the defective restoration was removed, the old restoration surface were sandblasted, and the tooth and restoration surfaces were coditoned with acid, then silane applied, next adhesive then new repair composite was added to repair the old restoration and restore the carious cavity.
  Arms: Sandblast-Silane-Adhesive treatment group

SUMMARY:
Research Problem : Advances in adhesive technologies have introduced several surface treatment concepts that enable the clinician to adhere resin-based composite restorations onto new composite materials. The service life of faulty direct composite restorations can be prolonged by composite repair wherein durable adhesion between old and new resin-based composite materials is established.

DETAILED DESCRIPTION:
Objectives : A randomized controlled clinical trial was designed to apply the latest results of evidence-based in vitro studies regarding resin-based repair protocol. The study aimed to assess the effect of adding silane coupling agent as a separate step on the clinical performance of repaired composite restorations and compare the results with those of using the usual etch and bond protocol.

Materials and Methods : 45 patients were recruited for this study from patients attending the restorative dentistry clinics for postgraduate students, Jordan University of Science and Technology. Each patient had at least two defected posterior composite restorations that are indicated for repair. With this selection, 116 restorations with localized anatomical deficiencies and/or secondary caries were randomly assigned into three groups according to the type of surface treatment each tooth will receive before the application of the new composite material (Filtek Z250,3M,USA). The teeth in the control group (n = 45): were treated with 37% phosphoric acid etching and conventional one step adhesive (Single Bond,3M,USA). In the Silane-Adhesive group (n = 26): teeth were treated with acid etching and silane coupling agent application (Bis-silane) prior to adhesive bond (Adper single bond). In the Sandblast-Silane-Adhesive group (n = 45): teeth were treated with intra-oral sandblasting and silane coupling agent application (Bis-silane) prior to (Adper Single Bond). The reason of repair, age of old restorations and the location of the restoration-repair interfaces were recorded for every failed restorations. Two examiners followed-up and evaluated the restoration quality after an average of 6 months using modified USPHS criteria. The results of clinical performance were assessed using Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Deciduous tooth
* Sustained dentin hypersensitivity
* Irreversible pulpitis , necrotic, or inadequately-treated endodontic teeth
* Grossly defective composite restorations that were indicated for replacement.
* Teeth with compromised periodontal status.
* Patients with poor oral hygiene

Exclusion Criteria:

* Patients older than 18 years.
* Asymptomatic restored premolars or molars.
* Vital or endodontically treated teeth
* Patients with localized, marginal, anatomical deficiencies and/or carious lesions adjacent to composite restorations or esthetically unpleasant restorations.
* Teeth with marginal gingivitis but healthy periodontium.
* Tooth in normal occlusion with antagonist and at least one adjacent tooth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the quality of the repaired restoration retention, colour match, marginal discoloration, marginal adaptation, anatomical form and surface roughness. | 2 years
  Clinical examination and evaluation of the restoration quality according to the United States Public Health Service (USPHS) criteria as Alpha, Bravo and Charlie. Alpha scores mean a better outcome and Charlie scores mean worse outcome.

SECONDARY OUTCOMES:
The presence of postoperative sensitivity. | 2 years.
  Patients record their sensitivity in treated teeth and score its intensity on visual analogue scale (VAS) which was divided into 10 digits from 0 to 10 where scores from 0 to less than 5 mean "bearable sesitivity" and scores from 5 to10 mean "unbearable sensitivy" outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zakereyya Albashaireh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
A consent has to be obtained from the faculty of graduate studies for sharing data as data form part of graduate students thesis.

REFERENCES:
- [Derived] Albashaireh ZSM, Maghaireh GA, Alsaafeen HN. Effects of silane coupling treatment on the clinical performance of direct repaired resin-based composite (RBC) restorations with or without prior surface sandblasting: A randomized controlled trial. J Dent. 2023 Dec;139:104740. doi: 10.1016/j.jdent.2023.104740. Epub 2023 Oct 8. PMID 37816489